CLINICAL TRIAL: NCT05025033
Title: Chemotherapy Combined With Apatinib and PD-1 Monoclonal Antibody for Second-line or Above Treatment of Advanced Gastric Cancer-A Prospective, Single-arm, Open, Phase II Study
Brief Title: Chemotherapy Combined With Apatinib and PD-1 Antibody
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJMUCH-GI-GC01
Record Dates: First submitted 2021-01-13; First posted 2021-08-27 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2021-01

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; second-line treatment; chemotherapy; Apatinib mesylate; immunotherapy; PD-1 antibody
MeSH Terms: conditions — Stomach Neoplasms | interventions — Paclitaxel; Irinotecan; apatinib; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 antibody combined with apatinib and chemotherapy (Experimental): PD-1 antibody: 200mg intravenous drip every 3 weeks; Apatinib: 250mg/day; Chemotherapy: Irinotecan: 150mg/m2, intravenous drip every 2 weeks, or Paclitaxel: 150mg/m2, intravenous drip once every 3 weeks.
  Interventions: Drug: PD-1 antibody, paclitaxel or irinotecan, Apatinib mesylate

INTERVENTIONS:
Drug: PD-1 antibody, paclitaxel or irinotecan, Apatinib mesylate — PD-1 antibody 200mg intravenous drip every 3 weeks; Apatinib 250mg/day; Chemotherapy: Irinotecan 150mg/m2, intravenous drip every 2 weeks, or Paclitaxel 150mg/m2, intravenous drip, once every 3 weeks.
  Other Names: PD-1 antibody, chemotherapy,Apatinib

SUMMARY:
The effective rate of second-line and later-line single-agent therapy for advanced gastric cancer is limited. This research plan aims to explore whether the combination of drugs can further improve the benefits of second-line and above therapies. Previous studies have shown that there is a significant synergistic effect between chemotherapy and PD-1 monoclonal antibody, or anti-angiogenic TKI drugs and PD-1 monoclonal antibody. This project is planned to be based on the classic chemotherapy drugs irinotecan or paclitaxel, combined with mesylate Apatinib and PD-1 monoclonal antibody, explore the effectiveness and safety of this three-drug combination regimen for the second-line and above treatment of advanced gastric cancer, in order to provide a better late-line treatment plan for patients with advanced gastric cancer.

DETAILED DESCRIPTION:
This study is a prospective, single-center, single-arm phase II clinical study, which aims to explore the efficacy of PD-1 antibody combined with apatinib combined with chemotherapy as a second-line and above regimen in the treatment of advanced gastric cancer.The enrolled patients were patients with advanced inoperable gastric cancer or gastroesophageal junction adenocarcinoma who had advanced first-line fluorouracil combined with platinum or advanced second-line paclitaxel and irinotecan, with an ECOG PS of 0-1. Treatment plan: PD-1 antibody: 200mg intravenous drip every 3 weeks; Apatinib 250mg/day; Chemotherapy: Irinotecan 150mg/m2, intravenous drip every 2 weeks, or Paclitaxel 150mg/m2, intravenous drip, once every 3 weeks. An imaging evaluation is performed every 6-8 weeks. Monitor blood routine, blood biochemistry, electrocardiogram, urine routine, thyroid function, heart function according to clinical routine, and record adverse events. Primary observational endpoints: objective effective rate (ORR), progression-free survival time (PFS), secondary observational endpoints: overall survival time (OS), disease control rate (DCR) and safety, and dynamic monitoring of serum biomolecular markers for exploration study .

ELIGIBILITY:
Inclusion Criteria:

Patient age ≥18 years old;

1. The ECOG score is 0-1 points;
2. Patients with locally advanced gastric cancer or GEJ adenocarcinoma who have been histologically confirmed, metastatic or unresectable;
3. Have received at least one systemic chemotherapy regimen in the past and have progressed; or have received adjuvant chemotherapy, but the disease has progressed or relapsed within 6 months after the end of the treatment; have not used any of the drug treatments in this study;
4. There are measurable lesions that meet the RECIST 1.1 standard;
5. It has sufficient organ and bone marrow function, and the laboratory examination meets the following requirements: a.HGB≥90g/L;b.NEUT≥1.5×109/L;c.PLT ≥100×109/L;d. BIL≤1.5 times the upper limit of normal (ULN);e. ALT and AST≤2.5×ULN; liver metastasis, then ALT and AST≤5×ULN;f. Endogenous creatinine clearance rate ≥50ml/min (Cockcroft-Gault formula);g. Urine routine is normal, or urine protein <(++), or 24-hour urine protein <1.0 g;
6. Normal blood coagulation, no active bleeding and thrombosis: a. International normalized ratio INR≤1.5;b. Partial thromboplastin time APTT≤1.5 ULN;
7. Women of childbearing age must undergo a negative pregnancy test (serum or urine) within 14 days before enrollment, and voluntarily use appropriate methods of contraception during the observation period and within 8 weeks after the last administration of the study drug; for men, it should be surgery Sterilize or agree to use appropriate methods of contraception during the observation period and within 8 weeks after the last administration of the study drug;
8. Estimated survival period ≥ 3 months;
9. The patient voluntarily joined the study and signed an informed consent form (ICF);Those who are expected to have good compliance can follow up the efficacy and adverse reactions as required by the protocol.

Exclusion Criteria:

1. Have received anti-angiogenesis drug therapy in the past;
2. Have received anti-PD-1 and anti-PD-L1 antibody drug therapy in the past;
3. Patients with high blood pressure who cannot be reduced to the normal range by antihypertensive drugs (systolic blood pressure>140 mmHg, diastolic blood pressure>90 mmHg), coronary heart disease above grade I, grade I arrhythmia (including QTc interval prolongation) Male>450 ms, female>470 ms) and grade I cardiac insufficiency;
4. There are many factors that affect oral drugs (such as inability to swallow and intestinal obstruction, etc.);
5. Allergic to the drugs in this program;
6. Patients with a clear gastrointestinal bleeding tendency, including the following conditions: local active ulcer lesions, and fecal occult blood (+ +) cannot be included in the group; patients with a history of melena and hematemesis within 1 month;
7. Patients with contraindications to apatinib: For patients with active bleeding, intestinal perforation, intestinal obstruction, within 30 days after major surgery, drug-uncontrollable hypertension, grade Ⅲ-Ⅳ cardiac insufficiency (NYHA standard), severe liver and kidney Patients with dysfunction (Grade 4); If you have immune system diseases, you need to use a daily dose of dexamethasone above 10mg;
8. According to the judgment of the investigator, patients with concomitant diseases that seriously endanger the safety of the patient or affect the completion of the study;
9. The researcher believes that it is not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
The Overall Response Rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  The proportion of CR and PR
Progression Free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Time from the start of treatment to the progression of the disease

SECONDARY OUTCOMES:
Overall survival | From date of randomization until the date of death from any cause or the last visit date, whichever came first, assessed up to 60 months
  Time from the start of treatment to the occurrence of death
Disease Control rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  The proportion of CR,PR and SD
adverse events | Until 3 months after the end of the treatment
  The incidence of various adverse events

OTHER OUTCOMES:
biomolecular markers | From the begaining of treatment, then every 2 months after treatment, until the last time after treatment， assessed up to 24 months
  Serum will be collected before medication and during each evaluation. Mass spectrometry or RNA sequencing technology will be used to detect the differences in the exosomal proteome and non-coding RNA group in the serum before medication. Screen out the group of exosomal protein/non-coding RNA components with obvious differences in the two groups of patients; and consider its biological function/signal pathway, and finally select 1-2 kinds of protein/non-coding RNA.

CONTACTS AND LOCATIONS:
Overall Officials: Ting Deng, MD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fuchs CS, Doi T, Jang RW, Muro K, Satoh T, Machado M, Sun W, Jalal SI, Shah MA, Metges JP, Garrido M, Golan T, Mandala M, Wainberg ZA, Catenacci DV, Ohtsu A, Shitara K, Geva R, Bleeker J, Ko AH, Ku G, Philip P, Enzinger PC, Bang YJ, Levitan D, Wang J, Rosales M, Dalal RP, Yoon HH. Safety and Efficacy of Pembrolizumab Monotherapy in Patients With Previously Treated Advanced Gastric and Gastroesophageal Junction Cancer: Phase 2 Clinical KEYNOTE-059 Trial. JAMA Oncol. 2018 May 10;4(5):e180013. doi: 10.1001/jamaoncol.2018.0013. Epub 2018 May 10. PMID 29543932
- [Background] Kang YK, Boku N, Satoh T, Ryu MH, Chao Y, Kato K, Chung HC, Chen JS, Muro K, Kang WK, Yeh KH, Yoshikawa T, Oh SC, Bai LY, Tamura T, Lee KW, Hamamoto Y, Kim JG, Chin K, Oh DY, Minashi K, Cho JY, Tsuda M, Chen LT. Nivolumab in patients with advanced gastric or gastro-oesophageal junction cancer refractory to, or intolerant of, at least two previous chemotherapy regimens (ONO-4538-12, ATTRACTION-2): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2017 Dec 2;390(10111):2461-2471. doi: 10.1016/S0140-6736(17)31827-5. Epub 2017 Oct 6. PMID 28993052
- [Background] Apetoh L, Ladoire S, Coukos G, Ghiringhelli F. Combining immunotherapy and anticancer agents: the right path to achieve cancer cure? Ann Oncol. 2015 Sep;26(9):1813-1823. doi: 10.1093/annonc/mdv209. Epub 2015 Apr 28. PMID 25922066
- [Background] Bang YJ, Kang YK, Catenacci DV, Muro K, Fuchs CS, Geva R, Hara H, Golan T, Garrido M, Jalal SI, Borg C, Doi T, Yoon HH, Savage MJ, Wang J, Dalal RP, Shah S, Wainberg ZA, Chung HC. Pembrolizumab alone or in combination with chemotherapy as first-line therapy for patients with advanced gastric or gastroesophageal junction adenocarcinoma: results from the phase II nonrandomized KEYNOTE-059 study. Gastric Cancer. 2019 Jul;22(4):828-837. doi: 10.1007/s10120-018-00909-5. Epub 2019 Mar 25. PMID 30911859
- [Background] Hughes PE, Caenepeel S, Wu LC. Targeted Therapy and Checkpoint Immunotherapy Combinations for the Treatment of Cancer. Trends Immunol. 2016 Jul;37(7):462-476. doi: 10.1016/j.it.2016.04.010. Epub 2016 May 20. PMID 27216414
- [Background] Kawazoe A, Fukuoka S, Nakamura Y, Kuboki Y, Wakabayashi M, Nomura S, Mikamoto Y, Shima H, Fujishiro N, Higuchi T, Sato A, Kuwata T, Shitara K. Lenvatinib plus pembrolizumab in patients with advanced gastric cancer in the first-line or second-line setting (EPOC1706): an open-label, single-arm, phase 2 trial. Lancet Oncol. 2020 Aug;21(8):1057-1065. doi: 10.1016/S1470-2045(20)30271-0. Epub 2020 Jun 23. PMID 32589866
- [Background] Xu J, Zhang Y, Jia R, Yue C, Chang L, Liu R, Zhang G, Zhao C, Zhang Y, Chen C, Wang Y, Yi X, Hu Z, Zou J, Wang Q. Anti-PD-1 Antibody SHR-1210 Combined with Apatinib for Advanced Hepatocellular Carcinoma, Gastric, or Esophagogastric Junction Cancer: An Open-label, Dose Escalation and Expansion Study. Clin Cancer Res. 2019 Jan 15;25(2):515-523. doi: 10.1158/1078-0432.CCR-18-2484. Epub 2018 Oct 22. PMID 30348638
- [Derived] Zhang L, Wang W, Ge S, Li H, Bai M, Duan J, Yang Y, Ning T, Liu R, Wang X, Ji Z, Wang F, Zhang H, Ba Y, Deng T. Sintilimab Plus Apatinib and Chemotherapy as Second-/Third-Line treatment for Advanced Gastric or Gastroesophageal Junction Adenocarcinoma: a prospective, Single-Arm, phase II trial. BMC Cancer. 2023 Mar 5;23(1):211. doi: 10.1186/s12885-023-10661-4. PMID 36872337

DOCUMENTS (1):
  • Informed Consent Form (2020-10-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT05025033/ICF_000.pdf